CLINICAL TRIAL: NCT00100776
Title: Efficacy of High Dose Olanzapine in a Controlled Fixed Dose-Response Trial for the Treatment of Schizophrenia and Schizoaffective Disorder
Brief Title: Efficacy of High Dose Olanzapine for the Treatment of Schizophrenia and Schizoaffective Disorder
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 8333; F1D-US-HGLF
Record Dates: First submitted 2005-01-06; First posted 2005-01-07 (Estimated); Last update posted 2007-01-26 (Estimated); Status verified 2007-01

CONDITIONS: Schizophrenia; Schizoaffective Disorder
MeSH Terms: conditions — Schizophrenia; Psychotic Disorders | interventions — Olanzapine

INTERVENTIONS:
Drug: Olanzapine

SUMMARY:
The purposes of this study are to assess the efficacy, safety, and side effects among doses approved by the Food and Drug Administration and higher (not FDA approved) doses of olanzapine in patients with schizophrenia or schizoaffective disorder.

ELIGIBILITY:
Inclusion Criteria:

* You must be 18 to 60 years old
* You must have been diagnosed with schizophrenia or schizoaffective disorder
* You must be able to visit the doctor's office 8 times over a 9 week period
* You must agree to participate with all tests and examinations that are required for this study

Exclusion Criteria:

* You are a woman and are pregnant or breastfeeding
* You presently have an acute or unstable medical illness
* You have a history of an allergic reaction to olanzapine
* You are taking medications that are not permitted in this study. Your physician will discuss these with you
* You have taken part in another clinical research trial within the last 30 days or you have received treatment with a drug in the last 30 days that has not received regulatory approval.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 600
Dates: Start 2003-09; Study Completion 2005-11

PRIMARY OUTCOMES:
The primary objective of this study is to assess the fixed dose response relationship for efficacy between standard and higher doses of olanzapine (10, 20, and 40 mg/day) in patients with schizophrenia or schizoaffective disorder.

SECONDARY OUTCOMES:
To assess the dose response efficacy of olanzapine in improving psychopathology of schizophrenia as measured by a mean change from baseline on the PANSS subscores and Clinical Global Impression-Severity(CGI-S) Scale as well as by the absolute score
of CGI-I (Improvement) Scale
To assess the efficacy of olanzapine doses between treatment arms (e.g. 10 mg/day versus 40 mg/day ) in improving the psychopathology of schizophrenia as measured by mean changed from baseline on the PANSS total and subscores and Clinical Global
Impression-Severity (CGI-S) Scale as well as by absolute score of CGI-I (Improvement) Scale
To assess the efficacy of olanzapine doses as measured by efficacy scales in patients who have successfully completed the 2 week titration period
To assess the efficacy of olanzapine doses within the standard range of 10 and 20 mg/day versus high dose 40 mg/day in improving the psychopathology of schizophrenia as measured by mean change from baseline on the PANSS total
To assess the response rate of olanzapine doses in improving the psychopathology of schizophrenia. Clinical response is defined as an improvement (reduction) of =>20% from baseline in the PANSS total score
To compare the time to response among all olanzapine treatment arms. Clinical response is defined as an improvement (reduction) of =>20% from baseline in the PANSS total score. In addition, the cumulative frequency distribution of differential
rates of response reduction in PANSS total score will be assessed at 8 weeks
To compare the dose response efficacy between all olanzapine treatment arms in improving depressive symptoms as measured by a mean change from baseline on the Montgomery-Asberg Depression Rating Scale (MADRS)
To assess the efficacy between all olanzapine treatment arms in improving patients' overall level of functioning and health-related quality of life as measured by the Global assessment of Functioning (GAF) and the Heinrich Carpenter
Quality of Life Scale (QLS)
To analyze steady-state olanzapine plasma concentrations following 10, 20, and 40 mg daily dosing and examine the associations between state plasma levels, efficacy, and safety measures
To assess the safety between treatment arms and the safety dose-response relationship between the olanzapine treatment groups as determined by:
Treatment-emergent adverse events,
ECG
Vital signs and fasting laboratory analytes (clinical chemistry, hematology, lipid panel, and prolactin)
Appetite as measured by the Eating Behavior Assessment
Extrapyramidal symptoms as measured by the Modified Simpson-Angus Scale, The Barnes Akathisia Rating Scale, and the Abnormal Involuntary Movement Scale (AIMS)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (33):
- United States (33):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Monday-Friday from 9:00 AM to 5:00 PM Eastern Time (UTC/GMT-5 hours, EST), or speak with your personal physician, Anaheim, California
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Monday-Friday from 9:00 AM to 5:00 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician, National City, California
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Monday-Friday from 9:00 AM to 5:00 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician, Orange, California
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Monday-Friday from 9:00 AM to 5:00 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician, Pasadena, California
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Monday-Friday from 9:00 AM to 5:00 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician, San Diego, California
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Monday-Friday from 9:00 AM to 5:00 PM Eastern Time (UTC/GMT-5 hours, EST), or speak with your personal physician, New Britain, Connecticut
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Monday-Friday from 9:00 AM to 5:00 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician, Washington D.C., District of Columbia
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Monday-Friday from 9:00 AM to 5:00 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician, Fort Lauderdale, Florida
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Monday-Friday from 9:00 AM to 5:00 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician, Hialeah, Florida
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Monday-Friday from 9:00 AM to 5:00 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician, Winter Park, Florida
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Monday-Friday from 9:00 AM to 5:00 PM Eastern Time (UTC/GMT-5 hours, EST), or speak with your personal physician, Augusta, Georgia
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Monday-Friday from 9:00 AM to 5:00 PM Eastern Time (UTC/GMT-5-hours, EST), or speak with your personal physician, Chicago, Illinois
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Monday-Friday from 9:00 AM to 5:00 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician, Granite City, Illinois
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Monday-Friday from 9:00 AM to 5:00 PM Eastern Time (UTC/GMT-5 hours, EST), or speak with your personal physician, Hoffman Estates, Illinois
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Monday-Friday from 9:00 AM to 5:00 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician, Lafayette, Indiana
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Monday-Friday from 9:00 AM to 5:00 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician, Minneapolis, Minnesota
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Monday-Friday from 9:00 AM to 5:00 PM Eastern Time (UTC/GMT-5 hours, EST), or speak with your personal physician, Las Vegas, Nevada
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Monday-Friday from 9:00 AM to 5:00 PM Eastern Time (UTC/GMT-5 hours, EST), or speak with your personal physician, Reno, Nevada
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Monday-Friday from 9:00 AM to 5:00 PM Eastern Time (UTC/GMT-5-hours, EST), or speak with your personal physician, Clementon, New Jersey
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Monday-Friday from 9:00 AM to 5:00 PM Eastern Time (UTC/GMT-5 hours, EST), or speak with your personal physician, Kenilworth, New Jersey
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Monday-Friday from 9:00 AM to 5:00 PM Eastern Time (UTC/GMT-5 hours, EST), or speak with your personal physician, New York, New York
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Monday-Friday from 9:00 AM to 5:00 PM Eastern Time (UTC/GMT-5 hours, EST), or speak with your personal physician, Olean, New York
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Monday-Friday from 9:00 AM to 5:00 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician, Orangeburg, New York
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Monday-Friday from 9:00 AM to 5:00 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician, Staten Island, New York
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Monday-Friday from 9:00 AM to 5:00 PM Eastern Time (UTC/GMT-5 hours, EST), or speak with your personal physician, Butner, North Carolina
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Monday-Friday from 9:00 AM to 5:00 PM Eastern Time (UTC/GMT-5 hours, EST), or speak with your personal physician, Raleigh, North Carolina
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Monday-Friday from 9:00 AM to 5:00 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician, Beachwood, Ohio
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Monday-Friday from 9:00 AM to 5:00 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician, Cleveland, Ohio
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Monday-Friday from 9:00 AM to 5:00 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician, Oklahoma City, Oklahoma
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Monday-Friday from 9:00 AM to 5:00 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician, Madison, Tennessee
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Monday-Friday from 9:00 AM to 5:00 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician, Austin, Texas
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Monday-Friday from 9:00 AM to 5:00 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician, Houston, Texas
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Monday-Friday from 9:00 AM to 5:00 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician, Tacoma, Washington

REFERENCES:
- [Derived] Lindenmayer JP, Liu-Seifert H, Kulkarni PM, Kinon BJ, Stauffer V, Edwards SE, Chen L, Adams DH, Ascher-Svanum H, Buckley PF, Citrome L, Volavka J. Medication nonadherence and treatment outcome in patients with schizophrenia or schizoaffective disorder with suboptimal prior response. J Clin Psychiatry. 2009 Jul;70(7):990-6. doi: 10.4088/JCP.08m04221. Epub 2009 Jun 2. PMID 19497244
- [Derived] Citrome L, Stauffer VL, Chen L, Kinon BJ, Kurtz DL, Jacobson JG, Bergstrom RF. Olanzapine plasma concentrations after treatment with 10, 20, and 40 mg/d in patients with schizophrenia: an analysis of correlations with efficacy, weight gain, and prolactin concentration. J Clin Psychopharmacol. 2009 Jun;29(3):278-83. doi: 10.1097/JCP.0b013e3181a289cb. PMID 19440083